CLINICAL TRIAL: NCT03324438
Title: Home Telemedicine to Optimize Health Outcomes in High-Risk Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 17-0004; DP3DK113363 (NIH)
Record Dates: First submitted 2017-08-21; First posted 2017-10-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: MOST methodology uses factorial designs and the hypotheses in Aim 1 will be tested through a 2x2 factorial experiment, a highly efficient experimental design despite several common misconceptions about sample size requirements and power. A 2x2 factorial experiment is NOT a 4-arm trial in which each condition is compared in turn to a control condition. In fact, factorial designs do not require a larger number of participants than other designs (e.g., RCT) and when used to address suitable research questions, they require fewer participants than other designs. Adding factors does not require a dramatic increase in sample size to maintain power. The number of arms is listed below as 4 as # of arms is required by the clinicaltrails.gov site; please refer above for a more accurate description of the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Home Telehealth T1D (CoYoT1-HR) (Active Comparator): Home Telehealth T1D (C2oYoT1-HR), standard of care delivered via Telehealth for high-risk youth
  Interventions: Behavioral: Home Telehealth T1D C2oYoT1-HR
- Personalized Adherence Feedback (Experimental): C2oYoT1-HR+Personalized Adherence Intervention
  Interventions: Behavioral: Personalized Adherence Feedback
- Personalized Behavioral Health (Experimental): C2oYoT1-HR+Personalized Behavioral Health
  Interventions: Behavioral: Personalized Behavioral Health
- C2oYoT1-HR + Adherence + Behavioral (Experimental): C2oYoT1-HR + both Personalized Adherence Feedback + Personalized Behavioral Health (C2oYoT1-HR + Adherence + Behavioral)
  Interventions: Behavioral: Home Telehealth T1D C2oYoT1-HR; Behavioral: Personalized Behavioral Health; Behavioral: Personalized Adherence Feedback

INTERVENTIONS:
Behavioral: Home Telehealth T1D C2oYoT1-HR — 1) assessment of physical and behavioral health characteristics associated with high-risk status; 2) delivery of home telehealth that incorporates: 2a) medical and behavioral health care delivered with the endocrinologist and behavioral health specialist working together with high-risk youth; 2b) personalized intervention to improve T1D adherence and T1D clinical health outcomes; 2c) personalized intervention to improve mental health comorbidities and T1D clinical health outcomes; and 3) an underused methodological approach for optimizing intervention components to be delivered at point of care.
  Other Names: C2oYoT1-HR
  Arms: C2oYoT1-HR + Adherence + Behavioral; Home Telehealth T1D (CoYoT1-HR)
Behavioral: Personalized Behavioral Health — 1) assessment of physical and behavioral health characteristics associated with high-risk status; 2) delivery of home telehealth that incorporates: 2a) medical and behavioral health care delivered with the endocrinologist and behavioral health specialist working together with high-risk youth; 2b) personalized intervention to improve T1D adherence and T1D clinical health outcomes; 2c) personalized intervention to improve mental health comorbidities and T1D clinical health outcomes; and 3) an underused methodological approach for optimizing intervention components to be delivered at point of care.
  Other Names: C2oYoT1-HR + Behavioral Health
  Arms: C2oYoT1-HR + Adherence + Behavioral; Personalized Behavioral Health
Behavioral: Personalized Adherence Feedback — 1) assessment of physical and behavioral health characteristics associated with high-risk status; 2) delivery of home telehealth that incorporates: 2a) medical and behavioral health care delivered with the endocrinologist and behavioral health specialist working together with high-risk youth; 2b) personalized intervention to improve T1D adherence and T1D clinical health outcomes; 2c) personalized intervention to improve mental health comorbidities and T1D clinical health outcomes; and 3) an underused methodological approach for optimizing intervention components to be delivered at point of care.
  Other Names: C2oYoT1-HR + Personalized Adherence Intervention
  Arms: C2oYoT1-HR + Adherence + Behavioral; Personalized Adherence Feedback

SUMMARY:
This study addresses the critical need for improving Type 1 Diabetes (T1D) health outcomes in high-risk youth (A1C=9-12%; ages 10-17 yrs) (AIC: glycated hemoglobin) where suboptimal glycemic control has severe acute and long-term complications with potentially life threatening consequences. Lack of regular contact with T1D care providers, continued T1D nonadherence, and suboptimal behavioral and mental health functioning compromises the physical health of youth with T1D and the ability of T1D teams to provide effective treatment. If the aims of this study are achieved, this study will change T1D care practices by providing high-risk youth with T1D, and their parents, medical and behavioral health support via home telehealth intervention. This has the potential to significantly change access to T1D care, decrease time spent in hyperglycemia, reduce the frequency of hospital admissions, and improve glycemic control. In addition, this study's use of Multiphase Optimization Strategy (MOST), a highly efficient experimental strategy to determine effective intervention components, should be generalizable to all individuals with T1D, leading to cost-effective, home telehealth intervention programs. Innovative aspects include: 1) assessment of physical and behavioral health characteristics associated with high-risk status; 2) delivery of home telehealth that incorporates: 2a) medical and behavioral health care delivered with the endocrinologist and behavioral health specialist working together with high-risk youth; 2b) personalized intervention to improve T1D adherence and T1D clinical health outcomes; 2c) personalized intervention to improve mental health comorbidities and T1D clinical health outcomes; and 3) an underused methodological approach for optimizing intervention components to be delivered at point of care.

DETAILED DESCRIPTION:
AIM 1: PHASE 1: Use Multiphasic Optimization Strategy (i.e., MOST), a highly efficient experimental strategy, to determine specific components for inclusion in an intervention to 1a) improve primary clinical outcomes of A1C and percentage of time spent in hyperglycemia and 1b) address secondary clinical outcomes by improving adherence and biological markers of complications in high-risk pediatric patients with T1D (A1C=9-12%) as part of 12-month personalized behavioral intervention delivered via in-person T1D clinic visits and home telemedicine.

MOST methodology uses factorial designs and the hypotheses in Aim 1 will be tested through a 2x2 factorial experiment, a highly efficient experimental design despite several common misconceptions about sample size requirements and power. A 2x2 factorial experiment is NOT a 4-arm trial in which each condition is compared in turn to a control condition. In fact, factorial designs do not require a larger number of participants than other designs (e.g., Randomized Controlled Trials (RCT)) and when used to address suitable research questions, they require fewer participants than other designs. Adding factors does not require a dramatic increase in sample size to maintain power.

H1: There will be a main effect of Personalized Adherence Intervention on percentage of A1C, time spent in hyperglycemia, adherence behaviors, and biological markers of complications.

H2: There will be a main effect of Personalized Behavioral Health Intervention on percentage of A1C, time spent in hyperglycemia, adherence behaviors, and biological markers of complications.

AIM 2: PHASE 2: Determine effectiveness of the intervention components on maintenance of A1C, percentage of time spent in hyperglycemia, adherence, and biological markers improvements throughout 6-month follow-up.

H1: Participants who are randomized to T1D medical appointments every 6 weeks will show better improvements in gains in A1C, percentage of time spent in hyperglycemia, adherence, and biological markers compared to those participants who revert to medical appointments occurring every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* youth age 10-17 years
* A1C=9-12%
* parent(s) of child with confirmed diagnosis of T1D
* T1D duration >1 year
* parent and child agree to participate in home telehealth sessions
* ability to use telehealth equipment (i.e., computer, tablet, smartphone with internet connectivity)

Exclusion Criteria:

* developmental disability or reading disorder that prevents understanding of the intervention materials
* non-English speaking adolescents
* those with severe psychological disorders
* prescribed and taking medications that increase blood glucoses
* not seen in T1D clinic within the past year; pregnant if female; situational concerns (e.g., active custody battle)
* type 2 diabetes

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control (A1C): Change from baseline and every 12 weeks up to 72 weeks (18 mo) | weeks 1, 12, 24, 36, 48, 72
  A1C will be measured in the central lab located within the Barbara Davis Center at Study Visits 1 (week 1), 5 (week 24) and 9 (week 48), and Follow-Up Visit 2 (week 72) or 4 (week 72) which correspond to in-person T1D visits. In addition, participants will be asked to complete A1C measurements at an outside, independent Certified Laboratory Improvement Amendments (CLIA) lab prior to home telehealth T1D Study Visits 3 (week 12) and 7 (week 36). The rationale for measurement at these study visits is that they occur every 3 months, which is the interval in which A1C is measured as standard of care. Change in A1c will be looked at from baseline every 3 months throughout the study.
Hyperglycemia - Change from baseline and every 12 weeks up to 72 weeks (18 mo) | weeks 1, 12, 24, 36, 48, 72
  Time spent in hyperglycemia - change will be looked at from baseline every 12 weeks throughout the study.
Pediatric Diabetes Quality of Life Scale - Change from baseline and every 12 weeks up to 72 weeks (18 mo) | weeks 1, 12, 24, 36, 48, 72
  The PDQ is a 20-question self-administered scale that evaluates and quantifies the quality of life as related to diabetes - change will be looked at from baseline every 3 months throughout the study.

SECONDARY OUTCOMES:
Adherence - Change from baseline and every 12 weeks up to 72 weeks (18 mo) | weeks 1, 12, 24, 36, 48, 72
  Objectively Measured Adherence, Self-Reported Adherence, Number of T1D Appointments Attended. - change will be looked at from baseline every 3 months throughout the study.
Psychosocial Measures - Change from baseline and every 24 weeks up to 72 weeks (18 mo) | weeks 1, 24, 48, 72
  Diabetes Family Conflict Scale (DFCS), Diabetes Family Responsibility Questionnaire (DFRQ), Hypoglycemia Fear Scale (HFS), Patient Health Questionnaire - 9 (PHQ-9), Problem Area in Diabetes Version (PAID), Puberty - change will be looked at from baseline every 3 months throughout the study.
Biological Markers of T1D Complications - Change from baseline and every 24 weeks up to 72 weeks (18 mo) | weeks 1, 24, 48, 72
  Urinary microalbumin, endothelial function - change will be looked at from baseline every 3 months throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Driscoll, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
no sharing will occur at this point.